CLINICAL TRIAL: NCT05525988
Title: Proximal Pole Scaphoid Reconstruction Using Proximal Hamate: Case-Series on A Novel Technique
Brief Title: Proximal Pole Scaphoid Reconstruction Using Proximal Hamate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD 38/2022_FWA 00017585
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Closed Fracture Scaphoid, Proximal Pole; A Proximal Pole of Scaphoid That is Deemed Unsalvageable
Keywords: Proximal Pole Scaphoid Reconstruction, Hemi-Hamate Graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemi-Hamate Graft for Proximal Pole Scaphoid Reconstruction (Experimental): [All participants enrolled in this study for proximal pole scaphoid reconstruction using the Hemi-Hamate autograft]
  Interventions: Procedure: Hemi-Hamate Transfer for Proximal Pole Scaphoid Reconstruction

INTERVENTIONS:
Procedure: Hemi-Hamate Transfer for Proximal Pole Scaphoid Reconstruction — Surgical Technique:
  The participants will be positioned in the supine decubitus on the surgical table with the operated upper limb put on a C-arm (Mobile fluoroscopy device) compatible surgical arm-board. After anesthesia, a pneumatic tourniquet will be placed with a cuff pressure raised to 250 mmHg, then the limb is draped in the regular sterile fashion. Through a dorsal approach to the wrist joint, the proximal pole of scaphoid bone will be assessed before resectioning for confirmation that it cannot be preserved. The hamate bone will be exposed through capsulotomy and the measurements of the resected scaphoid will be transferred. The harvested H-H autograft will be placed and fixed to the distal scaphoid segment. Wound closure is then performed in layers in the usual fashion, and the wound will be covered by a sterile gauze, then a short-arm thumb spica splint will be put on.

SUMMARY:
Recently, A novel surgical technique was illustrated by Elhassan BT et al. in 2016 utilizing the Hemi-hamate autograft for the reconstruction of scaphoid bone proximal pole non-union with avascular necrosis.

The technique showed promising results but is still limited to case reports and anatomical studies

In this study, we aim to:

1. Evaluate the surgical technique steps and suggest any possible modifications to the original description of the technique.
2. Assessment of clinical outcomes of this novel technique in terms of; bone union rate, time to union, and wrist function.
3. Report any complications of the usage of the proximal hamate for the proximal pole of the scaphoid reconstruction.

DETAILED DESCRIPTION:
Almost 70 percent of all carpal bone fractures occur in the scaphoid bone, with an overall incidence of 12 per 100,000 of the general population. About 20 percent of scaphoid bone fractures are in the proximal third of the scaphoid, where the rates of ischemia were reported to be as high as 100 percent.

The risk of avascular necrosis (AVN) and/or non-union that in due course end in arthrosis with the fractures involving the proximal pole of the scaphoid is high and represents a challenging surgical problem, and even more challenging when the proximal pole is fragmented.

Several techniques were described for the surgical management of non-union of the proximal pole of scaphoid, including non-vascularised and vascularized bone grafts, each has characteristic pros and cons. Drawbacks with all of these techniques included donor-site morbidity and/or the requirement of microvascular skill in the case of a vascularized bone graft.

The Hemi-Hamate graft is the closest anatomically and histologically to the scaphoid compared to the rib costochondral and the medial femoral condyle grafts. The proximal part of the hamate has an analogous sizing and morphology to the proximal pole of the scaphoid bone. Both have a similar depth (palmar-dorsal breadth), width (radial-ulnar breadth), and sagittal radius of curvature.

Osteotomized proximal hamate with a maximum graft length at a level proximal to the hamulus distally did not adversely affect the lunate-capitate or the scaphoid-lunate kinematics during the wrist joint flexion-extension and the radial-ulnar deviation.

Since the technique was first described in 2016 only a single case-report study existed in the literature regarding the H-H autograft. Elhassan BT et al. reported that at 3.5-years follow-up the patient was free-pain, the wrist range of motion improved significantly and the Mayo wrist score was 90 which is coherent to an excellent outcome and, no symptoms of midcarpal instability were detected during 3.5-years follow-up.

The first case series published in the literature regarding the use of the Hemi-Hamate autograft was published by Saruhan S et al. in 2021; the study had a limited number of participants (4 cases) and, it was a retrospective study. In these four cases, the union was achieved, the pain was decreased, and there were no signs of donor-site morbidity at the final follow-up.

All probable complications have not been elucidated yet given the infancy stage of the technique description. Therefore, we decided to conduct a prospective case series study to report the outcomes of this newly developed promising technique and outline any possible drawbacks.

The investigators believe that this study will add significantly to the orthopedic literature given the infancy stage of this technique description.

Objectives:

1. Evaluate the surgical technique steps and suggest any possible modifications to the original description of the technique.
2. Assessment of clinical outcomes of this novel technique in terms of; bone union rate, time to union, and wrist function.
3. Report any complications of the usage of the proximal hamate for the proximal pole of the scaphoid reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Multifragmentary fracture of the proximal pole of scaphoid where fragments cannot be fixated.
* Participants with small and poor-quality proximal pole scaphoid bone fracture after the failure of a previous surgical fixation or bone grafting.

Exclusion Criteria:

* Proximal hamate arthrosis.
* Preexisting midcarpal instability.
* Arthritis at the radioscaphoid joint.
* Large hamate bone (Hamate radial-ulnar breadth greater than 1 cm in a participant with scaphoid bone radial-ulnar breadth less than 1 cm and palmar-dorsal breadth of less than 1.6 cm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Union Rate | 6 months postoperatively
  Reaching 50 percent graft union at the fracture site by Computed Tomography (CT) utilizing 1 mm thin cuts along the scaphoid long axis. [Done at the 6-week post-operative clinic visit to assess for the bone union and will be performed in monthly intervals till the bony union.]

SECONDARY OUTCOMES:
Time to Union | A 6 months postoperatively
  The time needed for the graft to reach 50 percent union at the fracture site by Computed Tomography (CT) utilizing 1 mm thin cuts along the scaphoid long axis. [Done at the 6-week post-operative clinic visit to assess for the bone union and will be performed in monthly intervals till the bony union.]
Complications | Intraoperatively to 1-year postoperatively
  Graft failure, malposition, malunion, delayed union, persistent non-union, carpal instability, and arthritis, as well as excessive scarring and complex regional pain syndrome, are all theoretically possible complications of this procedure.

OTHER OUTCOMES:
Range of Motion (ROM) of the Wrist | Preoperatively and 1-year postoperatively
  Evaluated by recording the (ROM) of the operated wrist using a goniometer
Mayo Wrist Score (MWS) | Preoperatively and 1-year postoperatively
  The Modified Mayo Wrist Score requires both patient and physician participation in order to assess pain, the active flexion/extension arc (in comparison with the contralateral side), grip strength (in comparison with the contralateral side), and the ability to return to regular employment or activities. Scores range from 0 to 100 with a score of 0 indicating a worse wrist condition and 100 indicating a better wrist condition.
The Patient Rated Wrist Evaluation (PRWE) sore | Preoperatively and 1-year postoperatively
  The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. The PRWE allows patients to rate their levels of wrist pain and disability from 0 to 10, and consists of 2 subscales:
  1. PAIN subscale (0 = no pain, 10 = worst ever)
     Pain - 5 items [Pain Score = Sum of the 5 pain items (out of 50)]
  2. FUNCTION subscale (0 = no difficulty, 10 = unable to do)
  Specific activities (6 items) and Usual activities (4 items) [Function Score = Sum of the 10 function items, Divided by 2 (out of 50)]
  Computing the Total Score: Total Score = Sum of pain + function scores
  Interpretation: Higher score indicates more pain and functional disability (e.g., 0 = no disability).
The Disabilities of the Arm, Shoulder and Hand (DASH) Score | Preoperatively and 1-year postoperatively
  The DASH is a 30-item self-reported questionnaire in which the response options are presented as 5-point Likert scales. Scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mohamed Ashraf Abdelfatah Rabie, Orthopedic Surgery Specialist,, Principal Investigator — Ain Shams University; Ayman Ibrahim Fathy Aly Hewaidy, Professor of Orthopedic Surgery,, Study Chair — Faculty of Medicine, Ain Shams University; Ahmed Naeem Atiyya Aly, Professor of Orthopedic Surgery,, Study Director — Faculty of Medicine, Ain Shams University; Amr Mostafa Mohamed Aly, Assistant Professor of Orthopedic Surgery,, Study Director — Faculty of Medicine, Ain Shams University; Ramy Ahmed Aly Soliman, Lecturer of Orthopedic Surgery,, Study Director — Faculty of Medicine, Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Greater Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chambers SB, Suh N. Proximal Hamate Autograft for Scaphoid Fractures: Surgical Anatomy and Technique. In: Bhatia DN, Bain GI, Poehling GG, Graves BR, eds. Arthroscopy and Endoscopy of the Elbow, Wrist and Hand. Springer, Cham; 2022: 899-905. https://doi.org/10.1007/978-3-030-79423-1_98
- [Background] Elhassan B, Noureldin M, Kakar S. Proximal Scaphoid Pole Reconstruction Utilizing Ipsilateral Proximal Hamate Autograft. Hand (N Y). 2016 Dec;11(4):495-499. doi: 10.1177/1558944716628497. Epub 2016 Mar 3. PMID 28149221
- [Background] Chan AHW, Elhassan BT, Suh N. The Use of the Proximal Hamate as an Autograft for Proximal Pole Scaphoid Fractures: Clinical Outcomes and Biomechanical Implications. Hand Clin. 2019 Aug;35(3):287-294. doi: 10.1016/j.hcl.2019.03.007. Epub 2019 May 11. PMID 31178087
- [Background] Saruhan S, Savran A, Yildiz M, Sener M. Reconstruction of proximal pole scaphoid non-union with avascular necrosis using proximal hamate: A four-case series. Hand Surg Rehabil. 2021 Dec;40(6):744-748. doi: 10.1016/j.hansur.2021.07.003. Epub 2021 Jul 16. PMID 34274497
- [Background] Wang DY, Li X, Shen ZC, Gu PL, Pei YR, Zeng G, Leng HJ, Zhang WG. [Three-dimensional architecture of intraosseous vascular anatomy of the hamate: a micro-computed tomography study]. Beijing Da Xue Xue Bao Yi Xue Ban. 2018 Apr 18;50(2):245-248. Chinese. PMID 29643522
- [Background] Wu K, Padmore C, Lalone E, Suh N. An Anthropometric Assessment of the Proximal Hamate Autograft for Scaphoid Proximal Pole Reconstruction. J Hand Surg Am. 2019 Jan;44(1):60.e1-60.e8. doi: 10.1016/j.jhsa.2018.04.021. Epub 2018 Jun 20. PMID 29934078
- [Background] Kakar S, Greene RM, Hewett T, Thoreson AR, Hooke AW, Elhassan BT. The Effect of Proximal Hamate Osteotomy on Carpal Kinematics for Reconstruction of Proximal Pole Scaphoid Nonunion With Avascular Necrosis. Hand (N Y). 2020 May;15(3):371-377. doi: 10.1177/1558944718793175. Epub 2018 Aug 20. PMID 30124083
- [Background] Sollaccio DR, Navo P, Ghiassi A, Orr CM, Patel BA, Lewton KL. Evaluation of Articular Surface Similarity of Hemi-Hamate Grafts and Proximal Middle Phalanx Morphology: A 3D Geometric Morphometric Approach. J Hand Surg Am. 2019 Feb;44(2):121-128. doi: 10.1016/j.jhsa.2018.06.008. Epub 2018 Jul 14. PMID 30017649
- [Background] Kakar S, Greene RM, Elhassan BT, Holmes DR 3rd. Topographical Analysis of the Hamate for Proximal Pole Scaphoid Nonunion Reconstruction. J Hand Surg Am. 2020 Jan;45(1):69.e1-69.e7. doi: 10.1016/j.jhsa.2019.05.013. Epub 2019 Jul 9. PMID 31300229
- [Background] Thayer MK, Bluth B, Huang JI. A Morphometric Analysis of Hamate Autograft for Proximal Scaphoid Reconstruction. J Wrist Surg. 2021 Jun;10(3):268-271. doi: 10.1055/s-0041-1726404. Epub 2021 Apr 14. PMID 34109073
- [Background] Robinson PG, Duckworth AD, Campbell DA. Acute Fractures in Sport: Wrist. In: Robertson GAJ, Maffulli N, eds. Fractures in Sport. Springer, Cham; 2021:155-174. https://doi.org/10.1007/978-3-030-72036-0_11
- [Background] Segalman KA, Graham TJ. Scaphoid Proximal Pole fractures and Nonunions. J. Am. Soc. Surg. Hand. 2004;4(4): 233-249. doi:10.1016/j.jassh.2004.09.008
- [Background] Gillis JA, Elhassan BT, Kakar S. Hamate to Scaphoid Transfer for Nonreconstructable Proximal Pole Scaphoid Fractures. In: Geissler WB, ed. Wrist and Elbow Arthroscopy with Selected Open Procedures. Springer, Cham; 2022: 555-559. https://doi.org/10.1007/978-3-030-78881-0_44